CLINICAL TRIAL: NCT06958458
Title: Empowering Mothers With Hospitalized Infants in the Neonatal Intensive Care Unit Through Integrated Care: A Randomized Controlled Trial
Brief Title: Empowering Mothers in the NICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Emel AVÇİN, Lecturer Dr, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Emel A. Family Integrated Care
Record Dates: First submitted 2025-04-18; First posted 2025-05-06 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Mothers; Premature; Empowerment
Keywords: Empowerment; Neonatal; Premature; Mothers; Nursing
MeSH Terms: conditions — Premature Birth; Empowerment

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial (RCT) designed to evaluate the effectiveness of an intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mother Integrated Care Group (Experimental): Mothers whose infants are admitted to the NICU will be contacted within the first 72 hours. Pre-test data (Information Form, Maternal Attachment Scale, and Parental Stressor Scale: Neonatal Intensive Care Unit) will be collected, and education will be planned through a face-to-face interview.
  After meeting with the mother and administering the pre-test, the training date will be scheduled together with the researchers.
  The training, which consists of four steps, is planned to be conducted with a two-day interval between each session.
  The practices will be demonstrated on mannequins and supported by a PowerPoint presentation and visual materials. A booklet prepared specifically for the mothers will also be distributed.
  After the training steps are completed, mothers will be encouraged to participate in their infant's care in cooperation with the NICU team.
  One day before discharge and one week after discharge, questionnaire forms will be administered via WhatsApp.
  Interventions: Behavioral: Mother Integrated Care
- Control group (No Intervention): Mothers in this group will receive standard unit care and education. Data collection procedures will be the same as those used in the intervention group. The mother will be contacted within the first 72 hours of admission to the unit, and pre-test data will be collected. One day before discharge and one week after discharge, questionnaire forms will be administered via WhatsApp.

INTERVENTIONS:
Behavioral: Mother Integrated Care — In order to empower mothers whose premature infants have been hospitalized in the neonatal intensive care unit (NICU) for at least three days, a four-step neonatal care training program will be provided. Through the empowerment of the mother, the empowerment of the family will also be supported. The family will no longer be considered as visitors but will be involved in the infant's care in the NICU as parents. Data collection forms will be completed before the training begins, one day prior to discharge, and one week after discharge.
  Arms: Mother Integrated Care Group

SUMMARY:
Family Integrated Care is designed to eliminate the barriers between parents and their infants in the NICU by involving parents of premature infants in their care. Parents are integrated into both the healthcare team and the care of their infant. Through this approach, parents are informed about how they can contribute to their infant's overall development, including neurological and sensory development, motor and behavioral progress, as well as practices such as touch, bonding, skin-to-skin contact, breastfeeding, and increasing breast milk production. They are also educated on general hygiene and care tasks such as diaper changing and body cleaning. This model places importance on the protection and enhancement of both the physical and psychological well-being of the parent and the infant. During this process, parents move beyond being mere "visitors" in the unit to becoming active "participants" and members of the care team. Family integrated care aims to support parents in becoming the primary caregivers for their infants, both during hospitalization and after discharge. This model not only provides education and counseling but also supports the family's comprehensive involvement in the infant's care.

ELIGIBILITY:
Inclusion Criteria:

* The newborn must be premature (gestational age >28 and <34 weeks),
* The infant must be admitted to the NICU and hospitalized for at least 3 days,
* The mother must be open to communication and cooperation,
* The mother must voluntarily agree to participate in the study,
* The mother must be literate,
* The mother must be able to speak and understand Turkish,
* The mother must be primiparous and experiencing motherhood for the first time,
* The mother must be over 18 years of age,
* Mothers in the intervention group must be present in the hospital for an average of 6-8 hours per day.

Exclusion Criteria:

* The newborn has a congenital anomaly (e.g., craniofacial anomalies such as cleft palate, cleft lip, or facial muscle paralysis),
* The newborn has a diagnosed gastrointestinal, neurological, or genetic disorder (e.g., necrotizing enterocolitis, hydrocephalus, Down syndrome, omphalocele, gastroschisis, short bowel syndrome, or other diseases),
* The newborn has a congenital heart defect requiring surgical intervention,
* The mother has a diagnosed psychiatric illness,
* The mother and/or father do not wish to participate in the study.

Withdrawal Criteria:

* The mother does not attend the training sessions during the study period,
* The mother fails to maintain cooperation throughout the study,
* The newborn is transferred to another healthcare center for any reason,
* The mother wishes to withdraw from the study,
* The newborn is diagnosed with a chronic illness during the study process.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — It will be conducted with mothers who have premature infants in the neonatal intensive care unit (NICU).
Enrollment: 54 (Estimated)
Dates: Start 2025-08-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Parental Stress in the Neonatal Intensive Care Unit | The mother will be asked to complete the scale form within the first 72 hours of admission to the unit, one day before discharge, and one week after discharge.
  The Parental Stressor Scale: Neonatal Intensive Care Unit (PSS:NICU) will be used to assess the level of parental perception of stressors arising from the physical and psychosocial environment of the intensive care unit. The scale consists of 34 items across three dimensions: Sights and Sounds, Infant Appearance and Behavior, and Parental Role Alteration. Higher scores on the scale indicate higher levels of parental stress (minimum: 0, maximum: 170).
Maternal Attachment | The mother will be asked to complete the scale form within the first 72 hours of admission to the unit, one day before discharge, and one week after discharge.
  The Maternal Attachment Scale consists of 26 items. The total score can range from 26 to 104. A higher score indicates a higher level of maternal attachment.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL AVÇİN, Doctor, Principal Investigator — University of Yalova
Locations (1):
- Yalova University, Yalova, Turkey (Türkiye)